CLINICAL TRIAL: NCT04405999
Title: Prevention of Infection and Incidence of COVID-19 in Medical Personnel Assisting Patients With New Coronavirus Disease: a Randomised Controlled Trial
Brief Title: Prevention of Infection and Incidence of COVID-19 in Medical Personnel Assisting Patients With New Coronavirus Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 05-20-02-С
Record Dates: First submitted 2020-05-18; First posted 2020-05-28 (Actual); Results first posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-03

CONDITIONS: Increased Risk of SARS-CoV-2 Infection
MeSH Terms: interventions — Bromhexine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bromhexine hydrochloride Group (Experimental): medical personnel at risk for COVID-19 infection with oral administration of Bromhexine hydrochloride
  Interventions: Drug: Bromhexine Hydrochloride
- Control Group (No Intervention): medical personnel at risk for COVID-19 infection without oral administration of Bromhexine hydrochloride

INTERVENTIONS:
Drug: Bromhexine Hydrochloride — Medical personnel at risk for COVID-19 infection will receive study medication for 14 days
  Arms: Bromhexine hydrochloride Group

SUMMARY:
This is a randomized controlled trial of the efficacy and safety evaluation of oral administration of Bromhexine hydrochloride for the prevention of SARS-CoV-2 infection and COVID-19 disease in medical personnel assisting patients with a new coronavirus disease

DETAILED DESCRIPTION:
This study aims to evaluate the oral administration of Bromhexine hydrochloride for the prevention of SARS-CoV-2 infection and COVID-19 disease in medical personnel assisting patients with a new coronavirus disease. The aim of the study is to determine the preventive role of this drug in the framework of reducing the incidence of coronavirus infection in risk groups (medical personnel). Several studies show, that the acute respiratory syndrome coronavirus SARS-CoV uses endosomal cysteine proteases cathepsin B and L (CatB/L) and the transmembrane protease serine type 2 (TMPRSS2) for the priming of the viral S-protein. The new coronavirus SARS-CoV-2 penetrates into alveolar epithelial type two cells through a similar mechanism. In detail, viral S-protein binds to pneumocyte angiotensin-converting enzyme 2 (ACE2) and then undergoes cleaving by TMPRSS2 in S1- and S2-subunits. This leads to the release of a fusion peptide, which allows the virus to enter the cell via endocytosis. Therefore, the protease TMPRSS2 can serve as a target for pharmacological agents to prevent the penetration of the SARS-CoV-2 into the cell. Bromhexine blocks the TMPRSS2 ability to activate a zymogen precursor of tissue plasminogen activator in vitro. Interestingly, TMPRSS2 is blocked by much lower concentrations then required to inactivate other proteases in the cell culture. However, these data cannot be simply extended to the clinical practice: whether the concentration of bromhexine in the lung tissue of properly treated patients would be enough to prevent the virus entry through the TMPRSS2-inactivation remains unclear. A randomized study in people at risk for coronavirus infection will clarify the role of Bromhexine hydrochloride as a prevention of this disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 years or more;
2. Negative test (PCR) for SARS-CoV-2 infection;
3. The absence of clinical manifestations of a respiratory infection;
4. Contact with patients with laboratory and / or clinically confirmed SARS-CoV-2 infection;
5. Signed informed consent to participate in the study.

Exclusion Criteria:

1. Intolerance to Bromhexine hydrochloride;
2. Work out of contact with SARS-CoV-2 infection;
3. Non-compliance with the rules for the use of personal protective equipment when working with SARS-CoV-2 infection (the rules for the use of personal protective equipment in accordance with the recommendations of the Ministry of Health of Russia and the internal orders of the Director General of Almazov NMRC, relevant to the dates of research);
4. Pregnancy and the period of breastfeeding;
5. Other circumstances that the researcher considers inappropriate to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2020-08-09 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evgeny Mikhaylov, MD, PhD, Study Director — Almazov National Medical Research Centre
Locations (1):
- Almazov National Medical Research Centre, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mikhaylov EN, Lyubimtseva TA, Vakhrushev AD, Stepanov D, Lebedev DS, Vasilieva EY, Konradi AO, Shlyakhto EV. Bromhexine Hydrochloride Prophylaxis of COVID-19 for Medical Personnel: A Randomized Open-Label Study. Interdiscip Perspect Infect Dis. 2022 Jan 29;2022:4693121. doi: 10.1155/2022/4693121. eCollection 2022. PMID 35103059

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was performed via the institution's electronic communication system and via personal contacts with healthcare providers. Following a general notification via an institutional electronic system, one hundred and fifty healthcare providers were contacted personally and 50 persons were included.
Pre-assignment Details: No subjects were excluded from the study before assignment to groups.
Groups:
- Treatment Group: medical personnel at risk for COVID-19 infection with oral administration of Bromhexine hydrochloride
  Bromhexine Hydrochloride: Medical personnel at risk for COVID-19 infection will receive study medication for 14 days
Period: Overall Study
Arm/Group | Treatment Group | Control Group
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bromhexine Hydrochloride Group | Control Group | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (6.9) | 39.5 (8.2) | 40.6 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 11 | 10 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 25 | 25 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Russia | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Negative Polymerase Chain Reaction (PCR)
Description: Number of Participants with Negative PCR of SARS-CoV-2 and The Absence of Clinical Manifestations of COVID-19 Infection in individuals taking Bromhexine hydrochloride 4 weeks after randomization.
Time Frame: 4 weeks after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 25 | 25
Participants | 2 | 7

2. Secondary Outcome: Number of Participants With Asymptomatic SARS-CoV-2 Infection
Description: Number of Participants with Asymptomatic SARS-CoV-2 Infection
Time Frame: 14 days after last contact
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 25 | 25
Participants | 2 | 2

3. Secondary Outcome: Number of Participants With Mild, Moderate and Severe COVID-19 Disease
Description: number of participants with mild, moderate and severe COVID-19 disease
Time Frame: 14 days after last contact
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 25 | 25
Participants | 0 | 5

4. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of Participants with Adverse Events
Time Frame: 14 days after last contact
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 25 | 25
Participants | 2 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 8 weeks.
Description: Overall number of participants affected by one or more Serious Adverse Events, for each arm/group.
Arm/Group | Bromhexine Hydrochloride Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 2/25 | 0/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bromhexine Hydrochloride Group (N=25) | Control Group (N=25)
Flash hot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — A short period of hot flashes at treatment initiation without sequelae. Treatment was not interrupted.
Acute cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Transient cough without sequelae. Drug treatment was not interrupted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-12): https://cdn.clinicaltrials.gov/large-docs/99/NCT04405999/Prot_SAP_000.pdf